CLINICAL TRIAL: NCT02888405
Title: Effects of Acute Dietary Changes on Estimates of Body Composition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None
Other Study IDs: 805223-2
Record Dates: First submitted 2016-08-19; First posted 2016-09-05 (Estimated); Last update posted 2016-09-05 (Estimated); Status verified 2016-08

CONDITIONS: Overweight
Keywords: Body Composition
MeSH Terms: conditions — Overweight | interventions — Diet, High-Protein Low-Carbohydrate; Diet, Carbohydrate-Restricted

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- High-carbohydrate diet (Experimental): Single day of 9 g/kg body weight consumption of carbohydrate. Isocaloric to very low-carbohydrate condition.
  Interventions: Other: High-carbohydrate diet
- Very low-carbohydrate diet (Experimental): Single day of 1 - 1.5 g/kg body weight consumption of carbohydrate. Isocaloric to high-carbohydrate condition.
  Interventions: Other: Low-carbohydrate diet

INTERVENTIONS:
Other: High-carbohydrate diet
  Arms: High-carbohydrate diet
Other: Low-carbohydrate diet
  Arms: Very low-carbohydrate diet

SUMMARY:
The present study sought to investigate the effects of acute dietary changes on estimates of body composition. Specifically, the impact of an acute high-carbohydrate diet (9 g/kg body weight of carbohydrate) and an acute very low-carbohydrate diet (1 - 1.5 g/kg body weight of carbohydrate) were examined.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy
* Recreationally active (>150 min/week of moderate or vigorous physical activity)
* Pre-menopausal with regularly occurring menstrual cycles over past 6 months (in females only)

Exclusion Criteria:

* Failure to meet inclusion criteria
* Commencement or cessation of taking the dietary supplement creatine within the past month
* Pregnant or may become pregnant during the study
* Known or suspected food allergy to any items used in study
* Presence of medical condition that could reasonably be negatively affected by participation

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2015-11; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Dual-energy X-ray Absorptiometry Output | 2 days
  Measures of lean soft tissue and fat mass obtained from dual-energy x-ray absorptiometry.
Bioelectrical Impedance Analysis Output | 2 days
  Measures of fat-free mass and fat mass obtained from bioelectrical impedance analysis.

IPD SHARING:
Plan to Share IPD: No